CLINICAL TRIAL: NCT00873015
Title: Safety and Pharmacokinetic Evaluation of Sodium Nitrite Injection for the Prevention of Post-Subarachnoid Hemorrhage Induced Vasospasm
Brief Title: Safety and Pharmacokinetic Evaluation of Nitrite for Prevention of Cerebral Vasospasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Pharmaceuticals (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14024; 1R44NS063485-01 (NIH)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Cerebral aneurysm; Subarachnoid hemorrhage; Nitrite
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm | interventions — Sodium Nitrite; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrite (Experimental): Continuous intravenous infusion of Sodium Nitrite
  Interventions: Drug: Sodium nitrite
- Vehicle control (Placebo Comparator): Continuous intravenous infusion of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Sodium nitrite — 14 day continuous infusion of one of 3 escalating doses of sodium nitrite: 32 nmol/min/kg, 48 nmol/min/kg, or 64 nmol/min/kg
  Other Names: Sodium Nitrite Injection NDC 60267-311-10
  Arms: Nitrite
Drug: Saline — 14 day continuous infusion of a vehicle control infusion
  Other Names: Sterile saline
  Arms: Vehicle control

SUMMARY:
The purpose of the study is to examine the safety of a 14 day infusion of sodium nitrite, and to study the pharmacokinetics of nitrite, during a 14 day infusion in patients with ruptured cerebral aneurysms.

DETAILED DESCRIPTION:
Intravenous sodium nitrite has been shown to prevent and to reverse cerebral vasospasm in a primate model of subarachnoid hemorrhage (SAH). This was a Phase IIA dose escalation study of sodium nitrite to determine its safety in patients with aneurysmal SAH and to establish its pharmacokinetics during a 14 day infusion.

Sodium nitrite was delivered intravenously for 14 days in 18 patients with SAH from a ruptured cerebral aneurysm using a dose escalation scheme in three cohorts of 6 patients each (3 nitrite, 3 saline), with a maximum dose of 64 nmol/min/kg. Sodium nitrite blood levels were frequently sampled and measured using mass spectroscopy and blood methemoglobin levels were continuously monitored using a pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

* Ruptured cerebral aneurysm

Exclusion Criteria:

* Pregnancy, sickle cell disease, G6PD deficiency, anticoagulant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Oldfield, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System Medical Center, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Oldfield EH, Loomba JJ, Monteith SJ, Crowley RW, Medel R, Gress DR, Kassell NF, Dumont AS, Sherman C. Safety and pharmacokinetics of sodium nitrite in patients with subarachnoid hemorrhage: a phase IIa study. J Neurosurg. 2013 Sep;119(3):634-41. doi: 10.3171/2013.3.JNS13266. Epub 2013 May 24. PMID 23706046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to University of Virginia Medical Center for the treatment of subarachnoid hemorrhage were screened for possible recruitment into this study.
Pre-assignment Details: Patients underwent neurosurgical repair of their subarachnoid hemorrhage prior to study recruitment and assignment.
Groups:
- Vehicle Control: Nitrite : 14 day continuous infusion of a vehicle control infusion
- Nitrite 32 Nmol/Min/kg: 14 day continuous infusion of sodium nitrite 32 nmol/min/kg
- Nitrite 48 Nmol/Min/kg: 14 day continuous infusion of sodium nitrite 48 nmol/min/kg
- Nitrite 64 Nmol/Min/kg: 14 day continuous infusion of sodium nitrite 64 nmol/min/kg
Period: Overall Study
Arm/Group | Vehicle Control | Nitrite 32 Nmol/Min/kg | Nitrite 48 Nmol/Min/kg | Nitrite 64 Nmol/Min/kg
Started | 9 | 4 | 3 | 3
Completed | 9 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 32 Nmol/Min/kg: Sodium nitrite : 14 day continuous infusion 32 nmol/min/kg
- 48 Nmol/Min/kg: Sodium nitrite: 14 day continuous infusion 48 nmol/min/kg
- 64 Nmol/Min/kg: Sodium nitrite: 14 day continuous infusion 64 nmol/min/kg
- Total: Total of all reporting groups
Arm/Group | 32 Nmol/Min/kg | Vehicle Control | 48 Nmol/Min/kg | 64 Nmol/Min/kg | Total
Number analyzed (Participants) | 4 | 9 | 3 | 3 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 3 | 3 | 18
  >=65 years | 0 | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (10) | 52 (18.3) | 50 (5) | 58 (7) | 51 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 2 | 13
  Male | 1 | 3 | 1 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 9 | 3 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Nitrite Concentration (Micromol/L)
Description: Samples for pharmacokinetic analysis were collected from subjects treated with sodium nitrite at -15, -5, 0, 10, 30, 60, and 90 minutes after starting nitrite infusion and then at 2, 4, 6, 8, 12, 24, and every 24 hours after starting nitrite infusion. The sample at the time of starting the infusion was considered to be the time 0 sample. On study day 14 additional blood samples were collected at 0, 10, 30, 60, and 90 minutes and at 2, 4, 6, 8, and 12 hours after stopping nitrite infusion. Blood samples were analyzed for nitrite levels using mass spectroscopy.
Time Frame: multiple time points up to the end of day 14
Population: Per protocol
Measure: Mean (Standard Deviation); unit: micromol/L
Groups:
- 64 Nmol/Min/kg: Sodium nitrite : 14 day continuous infusion of 64 nmol/min/kg
- 48 Nmol/Min/kg: Sodium nitrite : 14 day continuous infusion of 48 nmol/min/kg
- 32 Nmol/Min/kg: Sodium nitrite : 14 day continuous infusion of 32 nmol/min/kg
Arm/Group | 64 Nmol/Min/kg | 48 Nmol/Min/kg | 32 Nmol/Min/kg
Number analyzed (Participants) | 3 | 3 | 3
micromol/L | 4.2 (0.3) | 4.3 (0.4) | 2.6 (0.3)

2. Secondary Outcome: Safety of a 14 Day Infusion of Sodium Nitrite
Description: Development of methemoglobin > 5% or hypotension (systolic arterial blood pressure < 90 mm Hg for more than 15 minutes or < 80 mm Hg) during infusion of sodium nitrite
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Intravenous saline administration
Arm/Group | 64 Nmol/Min/kg | 48 Nmol/Min/kg | 32 Nmol/Min/kg | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 9
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Efficacy of 14 Day Infusion of Sodium Nitrite
Description: Development of vasospasm as documented by onset of neurologic symptoms and documentation of narrowing of vessel(s) on cerebral angiogram. Potential clinical vasospasm was evaluated as appropriate, based on the development of focal neurological deficits that suggested cerebral ischemia (such as hemiparesis and speech deficit) or global neurological deficit (altered level of consciousness) that could not be attributed to other etiologies (such as metabolic abnormalities, intracerebral hemorrhage, and hydrocephalus).
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Intravenous saline
Arm/Group | 64 Nmol/Min/kg | 48 Nmol/Min/kg | 32 Nmol/Min/kg | Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 9
Participants | 1 | 1 | 0 | 3

ADVERSE EVENTS:
Groups:
- Nitrite: Sodium nitrite : 14 day continuous infusion of one of 3 escalating doses of sodium nitrite: 32 nmol/min/kg, 48 nmol/min/kg, or 64 nmol/min/kg
Arm/Group | Nitrite | Vehicle Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrite (N=9) | Vehicle Control (N=9)
Abscess (Infections and infestations) | 0 (0) | 1 (1) — Abdominal abscess (secondary to percutaneous endoscopic gastrostomy tube dislodgement)
Death (Nervous system disorders) | 0 (0) | 1 (1) — Stroke progression (withdrawal of life support)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No